CLINICAL TRIAL: NCT05688280
Title: Intratumoral Injection of IP-001 Following Thermal Ablation in Patients With Advanced Solid Tumors. A Multicenter Phase 1b/2a Trial in Colorectal Cancer, Non-small Cell Lung Cancer, and Soft Tissue Sarcoma Patients
Brief Title: Intratumoral Injection of IP-001 Following Thermal Ablation in Patients With CRC, NSCLC, and STS
Acronym: INJECTABL-1
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immunophotonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP-IIO-622
Record Dates: First submitted 2022-12-22; First posted 2023-01-18 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Solid Tumor; Colon Cancer; Nonsmall Cell Lung Cancer; Soft Tissue Sarcoma
Keywords: Cancer; Anti-cancer drug or therapy; Advanced solid tumors; Intratumoral injection; IP-001; Thermal ablation; Phase lb/lla; Melanoma; Soft tissue sarcoma; Tumor ablation; Systemic immune response; Interventional immuno-oncology; Interventional oncology; Abscopal effect; T-cell stimulation
MeSH Terms: conditions — Neoplasm Metastasis; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Sarcoma; Neoplasms; Melanoma | interventions — N-dihydrogalactochitosan; Injections

STUDY DESIGN:
Intervention Model Description: Open-label study with 3 Cohorts
  * Cohort 1: 18 patients with Stage 3 or Stage 4 Colorectal Cancer (CRC)
  * Cohort 2: 17 patients with Stage 3 or Stage 4 Non-Small Cell Lung Cancer (NSCLC)
  * Cohort 3: 3 patients with Stage 3 or Stage 4 Soft Tissue Sarcoma (STS)
  There will be 3 study periods: a Pretreatment Period, a Treatment Period, and a Follow-up Period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Colorectal Cancer (CRC) (Experimental): Radiofrequency ablation (RFA) followed by an intratumoral injection of IP-001.
  Interventions: Drug: 1.0% IP-001 for Injection
- Non-Small Cell Lung Cancer (NSCLC) (Experimental): Radiofrequency ablation (RFA) followed by an intratumoral injection of IP-001.
  Interventions: Drug: 1.0% IP-001 for Injection
- Soft Tissue Sarcoma (STS) (Experimental): Radiofrequency ablation (RFA) followed by an intratumoral injection of IP-001.
  Interventions: Drug: 1.0% IP-001 for Injection

INTERVENTIONS:
Drug: 1.0% IP-001 for Injection — 4 mL 1.0% IP-001 for Injection following RFA every 6 weeks for up to 4 treatments.
  Other Names: IP-001

SUMMARY:
The goal of this clinical trial is to determine the safety and efficacy of IP-001 for intratumoral injection administration following thermal ablation of a solid tumor.

DETAILED DESCRIPTION:
The therapeutic approach taken by this clinical trial may offer patients a therapeutic benefit after failure of standard chemotherapy and immunotherapy.

Patients giving written informed consent will undergo screening during the Pretreatment Period to determine eligibility for trial entry. The Pretreatment Period will include collection and recording of medical history, concomitant medications, baseline symptoms, previous therapies, and baseline assessments. The patient's baseline tumor burden will be recorded with radiological assessments, along with analyzing location and size of tumors to identify and characterize target tumor(s) that will be treated and/or followed during the clinical trial.

If confirmed eligible for the study, the patient will advance into the Treatment Period. During the Treatment Period, patients will receive a routine radiofrequency ablation (RFA), followed by an injection of investigational product (IP-001 for Injection) into the tumor. Patients can be treated every 6 weeks for up to 4 treatments with RFA + IP-001 for Injection.

A patient will move to the 6-month Follow-up Period when the patient has completed 4 treatment cycles or if the decision is made that no subsequent treatments will be administered. During the Follow-up Period, there will be a Follow-up Visit every 6 weeks for 5 visits, at disease progression, or prior to the start of a new antineoplastic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Stage 3 or Stage 4 CRC, NSCLC, or STS who have failed, are ineligible, refused, or become intolerant to at least first line (but no more than 4 lines) of systemic therapy
2. Life expectancy of > 6 months. Only have lesions with the longest diameter of ≤ 5 cm.
3. Presence of at least one non-bone tumor lesion that is ablation-accessible, with a minimum size of 1.0 cm.
4. Measurable disease according to RECIST 1.1.
5. Age ≥ 18 years.
6. ECOG performance status 0-1.
7. Bone marrow function: neutrophil count ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, hemoglobin ≥ 90 g/L.
8. Adequate hematological function defined by white blood cell count ≥ 2.5 × 109/L with absolute neutrophil count ≥ 1.5 × 109/L, and hemoglobin ≥ 9 g/dL (transfusions allowed on study).
9. Adequate hepatic function defined by a total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range and aspartate transaminase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 × ULN for all patients, or for patients with documented metastatic disease to the liver and AST and ALT levels ≤ 5 × ULN. Patients with documented Gilbert disease are allowed if total bilirubin is less than 3 × ULN.
10. Adequate renal function defined by an estimated creatinine clearance ≥ 50 mL/min according to the Cockcroft-Gault formula (or local institutional standard method).
11. Men and women with childbearing potential agree to use effective contraception. Women of childbearing potential must have a negative pregnancy test (serum) before inclusion.

Exclusion Criteria:

1. Known allergic reaction to shellfish, crabs, crustaceans, or any trial components, used in trial treatment.
2. Malignant primary brain tumors or evidence of brain metastases or leptomeningeal disease.
3. Patients who have received chemotherapy, radiotherapy, immunotherapy, or concurrent or recent treatment with any other investigational agents within 21 days prior to treatment.
4. Patients who have not recovered to common terminology criteria for adverse events (CTCAE) Grade ≤ 1 from all side effects of prior therapies except for residual toxicities.
5. Patients with a history of malignancy, with the exception of non-melanoma skin cancers and in situ cancers.
6. Concomitant treatment with systemic corticosteroids (10 mg prednisolone or equivalent) or other immunosuppressive therapy.
7. Anti-coagulation therapies which cannot be stopped 24 hours prior to trial treatment.
8. Severe or uncontrolled cardiovascular disease (congestive heart failure New York Heart Association classification III or IV).
9. Documented HIV positive.
10. Active Hepatitis C or Hepatitis B Viral infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Up to 12 weeks
  The assessment of safety will be based on incidence of adverse events.

SECONDARY OUTCOMES:
Efficacy: Disease control according to Immune Response Evaluation Criteria in Solid Tumors for immune-based treatment (iRECIST) (iDC) | Up to 12 weeks
  An iDC is defined as any complete response (CR or iCR), partial response (PR or iPR), or stable disease (SD or iSD) for 12 weeks according to iRECIST achieved during the trial until disease progression according to iRECIST, death from any cause, or start of a subsequent anticancer treatment, whichever occurs first.
Efficacy: Disease control according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) (DC) | Up to 12 weeks
  A DC is defined as any complete response (CR), partial response (PR) or stable disease (SD) for 12 weeks from start of treatment according to RECIST 1.1 achieved during trial until disease progression according to iRECEST, death from any cause, or start of a subsequent anticancer treatment, whichever occurs first.
Efficacy: Objective response according to iRECIST (iOR) | Up to 12 weeks
  An iOR is defined as any complete response (CR or iCR) or partial response (PR or iPR) according to iRECIST achieved during the trial until disease progression according to iRECIST, death from any cause, or start of a subsequent anticancer treatment, whichever occurs first.
Efficacy: Duration of response according to iRECIST (iDOR) | Up to 12 weeks
  An iDOR is defined as the time from the first documentation of iOR until disease progression according to iRECIST (iPD) or death from any cause. iPD is defined as the time point of first iUPD without subsequent iSD, iPR or iCR before trial discontinuation.
Efficacy: Progression-free survival according to iRECIST (iPFS) | Up to 12 weeks
  An iPFS is defined as the time from treatment start until disease progression according to iRECIST (iPD) or death from any cause, whichever occurs first.
Efficacy: Objective response according to RECIST 1.1 (OR) | Up to 12 weeks
  An OR is defined as any complete response (CR) or partial response (PR) according to RECIST 1.1 achieved during trial until disease progression, death from any cause, or start of a subsequent anticancer treatment, whichever occurs first.
Efficacy: Duration of response according to RECIST 1.1 (DOR) | Up to 12 weeks
  A DOR is defined as the time from the first documentation of OR until disease progression according to RECIST 1.1, death from any cause, or start of a subsequent anticancer treatment, whichever occurs first.
Efficacy: Progression-free survival according to RECIST 1.1 (PFS) | Up to 12 weeks
  A PFS is defined as the time from treatment start until disease progression according to RECIST 1.1, or death from any cause, whichever occurs first.
Efficacy: Time to response according to iRECIST 1.1 (iTTR) | Up to 12 weeks
  An iTTR is defined as the time from start of trial treatment until iOR according to iRECIST achieved during the trial.
Efficacy: Time to response according to RECIST 1.1 (TTR) | Up to 12 weeks
  A TTR is defined as the time from treatment start until OR according to iRECIST achieved during the trial.
Efficacy: Disease-free survival (DFS) | Up to 12 weeks
  A DFS is defined as the time from start of treatment that the patient survives without any signs or symptoms of cancer or death from any cause, whichever occurs first.
Efficacy: Overall survival (OS) | Up to 12 weeks
  An OS is defined as the time from start of treatment until death from any cause.
Efficacy: OR of the injected lesions according to RECIST 1.1 | Up to 12 weeks
  An OR of the ablated and injected (treated) lesions will be assessed using RECIST 1.1.
Efficacy: OR of the non-injected lesions according to RECIST 1.1 | Up to 12 weeks
  An OR of the non-ablated and non-injected (untreated) lesions will be assessed using the RECIST 1.1 until disease progression according to RECIST 1.1, death from any cause, or start of a subsequent anticancer treatment, whichever occurs first.
Efficacy: iOR of the injected lesions according to iRECIST | Up to 12 weeks
  An iOR of the ablated and injected (treated) lesions will be assessed using the iRECIST until disease progression according to RECIST 1.1, death from any cause, or start of a subsequent anticancer treatment, whichever occurs first.
Efficacy: iOR of the non-injected lesions according to iRECIST | Up to 12 weeks
  An iOR of the non-ablated and non-injected (untreated) lesions will be assessed using the iRECIST until disease progression according to RECIST 1.1, death from any cause, or start of a subsequent anticancer treatment, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Jorger, MD, Principal Investigator — Cantonal Hospital of St. Gallen; Diane Beatty, PhD, Study Director — Immunophotonics, Inc.
Locations (16):
- United States (3):
  - Miami Cardiac & Vascular Institute, Coral Gables, Florida
  - University of Louisville Physicians, PSC, Louisville, Kentucky
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
- France (4):
  - Institut Bergonie, Bordeaux
  - Hospitalier Pitie-Salpetriere, Paris
  - Hôpital Foch, Suresnes
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Johann Wolfgang Goethe-Univresitat Frankfurt/Main, Frankfurt
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Munchen Klinik Bogenhausen, Munich
- Switzerland (4):
  - IOSI Ospedale San Giovanni Bellinzona, Bellinzona
  - Inselspital Universitatsspital, Bern, Bern
  - Kantonsspital Graubunden, Chur
  - Kantonsspital St. Gallen, Sankt Gallen
- United Kingdom (2):
  - University College London Hospitals, London
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No